CLINICAL TRIAL: NCT00834301
Title: An Open Label Trial to Evaluate the Effects of a Novel Renal Multivitamin on Inflammation and Other Biomarkers in Endstage Renal Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nephrian (Industry)
Responsible Party: Ray Chow, Ph.D., Nephrian Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N0801
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Hyperphosphatemia; Inflammation; Renal Disease
Keywords: End Stage Renal Disease; Inflammation
MeSH Terms: conditions — Hyperphosphatemia; Inflammation; Kidney Diseases; Kidney Failure, Chronic | interventions — Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Dietary Supplement: Oral Multivitamin

INTERVENTIONS:
Dietary Supplement: Oral Multivitamin — Oral Multivitamin

SUMMARY:
The purpose of the study is to determine whether an ingestion of a new renal multivitamin supplement can have a beneficial effect on bone and mineral adn inflammation issues related to patients on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease patients on dialysis for at least 90 days deemed to be at low risk by the investigator for being hospitalized or have concurrent infections
* Serum phosphorous level > 5 mg/dl
* Stable phosphate binder regimen for 2 week prior to enrollment
* Stable dose of Vitamin D for 4 weeks prior to enrollment
* Stable calcimimetic dose for 4 week prior to enrollment

Exclusion Criteria:

* patients who are pregnant
* patients who have pre existing thrombocytopenia defined as a platelet count of <100 x 109/L
* abnormal LFTs
* baseline CRP > 15 g/dl
* known sensitivity to any of the active ingredients
* patients who are currently enrolled in a clinical trial, or who have been in a clinical trial in the last six months
* are currently taking any immunosuppressive medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy and safety of a novel renal multivitamin on markers of bone and mineral metabolism in an ESRD population. | 8 weeks

SECONDARY OUTCOMES:
To assess the efficacy and safety of a novel renal multivitamin on markers of inflammation in an ESRD population | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ray Chow, PhD, Study Director — Nephrian
Locations (1):
- Simi Valley Dialysis Center, Simi Valley, California, United States